CLINICAL TRIAL: NCT03052335
Title: The Comparison of the Efficiency of Colon Capsule Endoscopy and Optical Colonoscopy in Patients With Positive Immunochemical Fecal Occult Blood Test
Brief Title: The Efficiency of Colon Capsule Endoscopy in Colon Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military University Hospital, Prague (Other)
Collaborators: Masaryk University (Other); Institute for Clinical and Experimental Medicine (Other Government); University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Stepan Suchanek, MD., Ph.D., Head of Department of Gastrointestinal Endoscopy, Military University Hospital, Prague
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-29614A
Record Dates: First submitted 2017-01-31; First posted 2017-02-14 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Colon Cancer
Keywords: colorectal cancer; screening; colon capsule; colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pillcam® COLON 2 Capsule and colonoscopy (Experimental): Persons with positive immunochemical fecal occult blood tests will be examined by second generation colon capsule endoscopy (CCE2) and optical colonoscopy afterwards.
  Interventions: Device: Pillcam® COLON 2 Capsule; Procedure: Colonoscopy

INTERVENTIONS:
Device: Pillcam® COLON 2 Capsule — The second generation of PillCam colon capsule endoscopy (CCE-2) is 11.6 mm × 31.5 mm in size and has two imagers, that each have a 172° angle of view, allowing for almost 360° visual coverage of the colon. CCE-2 has an adaptive frame rate from 4 to 35 images per second. This means that the camera is able to capture up to 35 pictures while in motion whereas 4 images per second are captured when it is virtually stationary. During the examination the patient wears a sensor array which is attached to the abdomen and a data recorder for storage of the information generated by the ingested capsule. After the examination the data are downloaded into the workstation and a video is generated.
Procedure: Colonoscopy — Optical colonoscopy is the standard method for evaluating the colon

SUMMARY:
Main objective is to improve colorectal cancer (CRC) screening programme in the Czech Republic and decrease the disease incidence and mortality. The secondary aim is to verify the effectiveness of incorporation of the new minimally invasive device in the prevention programme.

DETAILED DESCRIPTION:
Multicentre, multidisciplinary (3 gastroenterology units; biostatistics department; cooperation with general practitioners), prospective study is focused on examination of individuals with average colorectal cancer (CRC) risk (asymptomatic, age 50-75 years).

In years 2017 - 2019, there will be 230 persons with positive semi-quantitative immunochemical fecal occult blood tests (FIT; QuikRead, Orion Diagnostica Oy, Finland) with cut-off level 75 ng/ml involved. Every person will be examined by second generation colon capsule endoscopy (CCE2) and optical colonoscopy afterwards.

Main objective is to show that the negative predictive value (NPV) of the CCE2 applied in patients with positive FIT results is sufficient to include this method in the National CRC screening as filter test with aim to reduce the necessity of subsequent optical colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age 50 - 75 years
* asymptomatic (no enterorhagy, weight loss or anemia)
* signed informed consent with the study and with colonoscopy

Exclusion Criteria:

* CRC high-risk group patients

  * having first degree relatives diagnosed with colorectal cancer at age ˂ 60 years
  * FAP, HNPCC and other hereditary CRC syndromes probands
  * positive personal medical history of colorectal neoplasia (advanced adenomatous polyp, colorectal cancer)
* recent diagnostic, follow-up or preventive colonoscopy in ≤ 3 years (FOBT-positive colonoscopy, screening colonoscopy)
* colonoscopy contraindication
* severe acute inflammatory bowel disease
* severe comorbidities; likely non-compliance of the patient
* no informed consent signed (with the study and/or with colonoscopy)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of the CCE2 for large polyps (≥ 10 mm) | 1 day

SECONDARY OUTCOMES:
CCE2 accuracy for detection of advanced adenomas | 1 day
CCE2 accuracy for detection of colon cancer | 1 day
CCE2 and optical colonoscopy acceptance (special questionnaire) | 1 day
Cost-effectiveness analyses: cost reduction of preventive colonoscopies spared | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Suchanek, Study Director — Military University Hospital, Prague
Locations (1):
- Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided